CLINICAL TRIAL: NCT04392024
Title: Clinical Outcome of Extended-depth-of-focus Trifocal Intraocualr Lens (Triumf) Implantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, tae-young chung, Professor, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-12-020
Record Dates: First submitted 2020-05-15; First posted 2020-05-18 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Presbyopia
Keywords: Depth and focus
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Triumf (Other): Subjects who have cataract surgery with Triumf IOL
  Interventions: Device: Triumf

INTERVENTIONS:
Device: Triumf — Triumf is intraocular lens which offers multifocal vision by extended depth of focus and diffractive optics.

SUMMARY:
Clinical outcome of extended-depth-of-focus trifocal intraocualr lens (Triumf) implantation

ELIGIBILITY:
Inclusion Criteria:

1. Adult at the age of 21 or older at the time of the pre-operative examination and willing to have surgery on their 2nd eye within 7-28 days of their 1st eye
2. Age-related cataract
3. A patient with preoperative corneal astigmatism from IOL Master less than 1 diopters
4. A patient want presbyopia correction at the same time as cataract surgery
5. A patient has the visual potential of 20/25 or better in each eye after cataract removal and IOL implantation
6. Written informed consent to surgery and participation in the study

Exclusion Criteria:

1. Those with other diseases that can affect capsule stability such as pseudoexoliation syndrome, glaucoma, traumatic cataract
2. Pregnant woman and lactating woman
3. A patient with history of ocular trauma or ocular surgery (Intraocular surgery, refractive surgery, ocular surface surgery) in either eye
4. A patient with evidence of keratoconus or significant irregular astigmatism on pre-operative topography in either eye
5. If expectations for presbyopia correction are too high
6. Those who are not able to read and understand the informed consent (illiterate or foreigners)

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2020-01-29 (Actual); Primary Completion 2022-01-22 (Actual); Study Completion 2022-01-26 (Actual)

PRIMARY OUTCOMES:
Uncorrected distant visual acuity | 3 months
  Visual acuity at distant with bare eyes
Uncorrected near visual acuity | 3 months
  Visual acuity at near with bare eyes

SECONDARY OUTCOMES:
Contrast sensitivity | 3 months
  Ability to recognize figure or letter at different contrast environment
Quality of Vision | 3 months
  Degree of various symptoms associated with vision

CONTACTS AND LOCATIONS:
Overall Officials: Tae-Young Chung, PhD, Study Chair — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea